CLINICAL TRIAL: NCT03308201
Title: Study Evaluating Hemay022 in Combination With Endocrine Therapy In Subjects With ER Positive and HER2 Positive Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM022BC1C01
Record Dates: First submitted 2017-09-29; First posted 2017-10-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemay022 and Exemestane (Experimental): Part one: Hemay022 in combination with exemestane will be taken orally once daily. Planned dose escalation of Hemay022 will be 200mg, 300mg,400mg or 500mg daily for 28 days.
  Part two: Hemay022 in combination with exemestane will be taken in OTR dose until disease progression, intolerable toxicity or death.
  Interventions: Drug: Hemay022+exemestane
- Hemay022 and Letrozole (Experimental): Part two: Hemay022 in combination with letrozole will be taken in OTR dose until disease progression, intolerable toxicity or death.
  Interventions: Drug: Hemay022+letrozole
- Hemay022 and Fulvestrant (Experimental): Part two: Hemay022 in combination with fulvestrant will be taken in OTR dose until disease progression, intolerable toxicity or death.
  Interventions: Drug: Hemay022+ fulvestrant

INTERVENTIONS:
Drug: Hemay022+exemestane — Part one: Hemay022 tablets will be taken orally once daily in doses of 200mg, 300mg,400mg or 500mg for 28 days in combination with exemestane.
  Part two: Hemay022 tablets combination with exemestane.
  Arms: Hemay022 and Exemestane
Drug: Hemay022+letrozole — Part two: Hemay022 combination with letrozole.
  Arms: Hemay022 and Letrozole
Drug: Hemay022+ fulvestrant — Part two: Hemay022 combination with fulvestrant.
  Arms: Hemay022 and Fulvestrant

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Hemay022 combined with endocrine therapy in the treatment of ER and HER2-positive metastatic or advanced breast cancer, and to establish OTR (best tolerated regimen). The second purpose of this study is to evaluate the pharmacokinetics and efficacy of Hemay022 in combination with exemestane, and the safety of Hemay022 in combination with letrozole or fulvestrant.

The research will be divided into two parts. In the first part, 15 to 24 subjects will be enrolled to determine the safety and tolerability of combining Hemay022 with exemestane in patients with HER2-positive advanced breast cancer. The second part will enroll about 24-36 other subjects with ER and HER2-positive advanced breast cancer to better determine the tolerability and preliminary efficacy of Hemay022.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer subjects diagnosed by tumor histology;
2. Objective evidence shows that patients with metastasis or relapse who cannot be cured by standard treatment;
3. ER positive (≥1%) and HER2 over-expression (immunohistochemical IHC test 3+ and/or in situ hybridization ISH test positive), Post-menopausal female subjects who are suitable for exemestane as endocrine therapy ; Remarks: The expansion period is planned to include 6 subjects combined with letrozole and 6 subjects combined with fulvestrant in the 400mg dose group. Therefore, for this part of the subjects, the expansion period is included " Post-menopausal female subjects who are suitable for letrozole or fulvestrant as endocrine therapy";
4. Postmenopausal is defined as meeting any one of the following four conditions:

   * Past bilateral oophorectomy;
   * Age ≥60 years old;
   * Age <60 years old, natural menopause ≥12 months, in the past 1 year without chemotherapy, tamoxifen, toremifene or ovarian castration, the level of follicle stimulating hormone (FSH) and estradiol Within the postmenopausal range (use the reference range of the local laboratory).
   * Patients younger than 60 years old who are taking tamoxifen or toremifene, their FSH and estradiol levels are within the postmenopausal range (use the reference range of the local laboratory); Remarks: Premenopausal or perimenopausal women who do not meet the above-mentioned menopausal criteria can also be included in this study, but they must also receive zoladex ovarian suppression therapy. Ovarian suppression therapy has been started at least 14 days before the start of this program, and Must be continued during the treatment plan; For subjects whose postmenopausal status is difficult to judge, the investigator and medical personnel of the sponsor will determine whether to enter the group after discussion.
5. At least one evaluable tumor lesion (according to RECIST1.1) or only bone metastases;
6. ECOG Performance Status of 0-1;
7. The estimated survival time is more than 3 months;
8. Bone marrow function meets: ANC≥1.5×109/L, HB≥90 g/L (allowed for blood transfusion), PLT≥80×109/L. Liver function satisfies: ALT≤2.5×ULN, AST≤2.5×ULN, TBIL≤1.5×ULN (ALT≤5×ULN, AST≤5×ULN in patients with liver metastases); renal function satisfies: blood creatinine ≤1.5×ULN;
9. Subjects must give informed consent to the study before the study entry and voluntarily sign a written informed consent form;
10. The subject can communicate well with the investigator and can complete the research in accordance with the research regulations.

Exclusion criteria:

1. There are life-threatening visceral metastases, any central nervous system metastases or leptomeninges carcinomatosis;
2. Have received exemestane for breast cancer treatment (Note: If exemestane was previously used in the adjuvant treatment stage, and the drug has been stopped for ≥12 months before this enrollment, you can join the group); Remarks: For subjects who have been combined with letrozole in the extended phase, if they have received letrozole to treat breast cancer, they need to be excluded (if letrozole is used in the adjuvant treatment phase, and the drug has been stopped for ≥12 months before this enrollment , You can be included in the group); for subjects who have been combined with fulvestrant in the extended phase, if they have received fulvestrant for breast cancer, they need to be excluded.
3. The first-line endocrine therapy was used in the late stage, and the drug was stopped for less than 4 weeks;
4. Have received radiotherapy within 4 weeks prior to study;
5. Have received chemotherapy for advanced breast cancer> 2 lines (the subjects who have used chemotherapy drugs must have stopped the chemotherapy drugs for ≥ 4 weeks before being enrolled in this study);
6. Patients with parenteral nutrition; malabsorption syndrome; or any condition possibly affecting drug absorption or inability to tolerate oral medications;
7. Use of any drug that inhibits or induces hepatic metabolism of Hemay022 within 2 weeks prior to study and entire study duration, for example CYP3A4 strong inhibitors or strong inducers;
8. Patients who are known to have a history of allergies to Hemay022, exemestane or similar drugs (Note: For patients who are planning to combine letrozole or fulvestrant, if they are known to be allergic to letrozole or fulvestrant History cannot be included in this study);
9. Left ventricular ejection fraction (LVEF) <50％ as measured by echocardiogram or MUGA scan;
10. Positive blood for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening;
11. Complicated with ≥2 grade diarrhea or ≥2 grade nausea condition;
12. Active infection (ie, requiring intravenous antibiotic or antiviral agent);
13. Uncontrolled hypertension (systolic blood pressure> 150 mmHg, diastolic blood pressure> 100 mmHg after antihypertensive treatment);
14. Significant heart diseases, including ischemic heart disease (NYHA III-IV), history of myocardial infarction or uncontrolled angina within 6 months, occurrence congestive heart failure within 3 months;
15. Arrhythmias requiring treatment , including atrial fibrillation, supraventricular tachycardia ,ventricular tachycardia, ventricular fibrillation, or patients with coronary heart disease have symptoms requiring medicine treatment, myocardial infarction within 1 year, congestive heart failure (CHF);
16. Confirmed ECG abnormalities, including QTc (heart rate corrected according to Bazett formula or Fridericia formula) prolongation (≥450msec), QRS> 120ms;
17. History of hemorrhagic or thrombus events within 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, spontaneous tumor bleeding;
18. Have received other clinical trial treatments or other targeted drugs within 4 weeks before the study;
19. Major surgery or injury less than 4 weeks before the study;
20. Other chemotherapy, targeted therapy, hormone therapy, immunotherapy, radiotherapy (except symptomatic local radiotherapy) during the research;
21. Any other malignant cancer within 5 years with the exception of adequately treated cervical cancer in situ or basal and squamous cutaneous cell carcinomas;
22. History of alcohol or drug abuse;
23. Serious psychogenic illness;
24. Evidence of significant medical illness or abnormal laboratory finding that would make the subject inappropriate for this study by the investigator's judgment;
25. Subjects could not complete the study due to other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | from baseline until 4 weeks after the study day

SECONDARY OUTCOMES:
Objective response rate (complete response rate + partial response rate) according to RECIST v1.1 | At screening, every 8 weeks of treatment up to 18 months
Clinical benefit rate defined as percentage of patients with stable disease (SD) ≥ 6 months/partial response (PR)/complete response (CR). according to RECIST v1.1 | At screening, every 8 weeks of treatment up to 18 months
Progression Free Survival defined as the proportion of patients alive and without progression (according to RECIST v1.1 criteria) | 18 months after treatment initiation
Observed maximum concentration of Hemay022 and exemestane | 0, 0.5, 1, 2, 3, 4, 8, 12, 24 hours post-dose on day 1 and day 28
Time of maximum concentration of Hemay022 and exemestane | 0, 0.5, 1, 2, 3, 4, 8, 12, 24 hours post-dose on day 1 and day 28
Area under the plasma concentration versus time curve of Hemay022 and exemestane | 0, 0.5, 1, 2, 3, 4, 8, 12, 24 hours post-dose on day 1 and day 28
Trough Plasma Concentrations of Hemay022 and exemestane | pre-dose on day 14

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China